CLINICAL TRIAL: NCT02809378
Title: The Effects of Anesthetic Techniques and Palonosetron Administration on the Incidence of Postoperative Nausea and Vomiting in the Women Patients Undergoing Thyroidectomy
Brief Title: The Effects of Anesthetic Techniques and Palonosetron Administration on the Incidence of PONV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Collaborators: HK inno.N Corporation (Industry)
Responsible Party: Principal Investigator, DAE HEE KIM, Assistant Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MED-CT4-15-461
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: PONV; Palonosetron; Anesthesia
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Palonosetron; Sevoflurane; Remifentanil; Thiopental; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sevoflurane (Experimental): anesthesia induction with pentothal sodium (4-5 mg/kg), maintenance with sevoflurane(1.6-2.5 vol%)
  Interventions: Drug: sevoflurane; Drug: pentothal sodium
- sevoflurane, remifentanil, and propofol (Experimental): anesthesia induction and maintenance with remifentanil, propofol and sevoflurane(1.6-2.5 vol%)
  Interventions: Drug: sevoflurane; Drug: remifentanil; Drug: propofol
- Sevoflurane, remifentanil, propofol, and palonosetron (Experimental): anesthesia induction and maintenance with remifentanil, propofol and sevoflurane(1.6-2.5 vol%), and palonosetron 75 ug administration prior to anesthesia induction.
  Interventions: Drug: Palonosetron; Drug: sevoflurane; Drug: remifentanil; Drug: propofol

INTERVENTIONS:
Drug: Palonosetron — newly developed 5-HT3 antagonists with long half life (48 hrs) intravenous administration prior to anesthesia induction
  Arms: Sevoflurane, remifentanil, propofol, and palonosetron
Drug: sevoflurane — Inhalational anesthetics Halogenated.
Drug: remifentanil — ultra-short acting opioid anesthetics
  Arms: Sevoflurane, remifentanil, propofol, and palonosetron; sevoflurane, remifentanil, and propofol
Drug: pentothal sodium — intra-venous anesthetics for anesthesia induction
  Arms: Sevoflurane
Drug: propofol — intra-venous anesthetics for anesthesia induction and maintenance
  Arms: Sevoflurane, remifentanil, propofol, and palonosetron; sevoflurane, remifentanil, and propofol

SUMMARY:
The incidence of postoperative nausea and vomiting (PONV) after thyroidectomy have been shown to be relatively high compared other surgeries, with a reported incidence 65-75 %. PONV may increase patient discomfort, delay patient discharge, and increase the cost of patient care, the risk of postoperative bleeding which may potentially cause airway obstruction.

It is reported that the maintenance of anesthesia with propofol-remifentanil or sevoflurane-propofol-remifentanil decreased the incidence of PONV compared sevoflurane alone, but failed to demonstrate the decreased incidence of PONV in 6-24 hr postoperative period in patients undergoing thyroidectomy. Administration of Palonosetron, newly developed 5-HT3 antagonists with long half life (48 hrs) may decrease the incidence of PONV particularly during this period.

The purpose of this study was to evaluate and compare the incidence of PONV after thyroidectomy with three different anesthetic methods, sevoflurane or sevoflurane-propofol-remifentanil or sevoflurane-propofol-remifentanil-palonosetron in woman patients.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thyroidectomy euthyroid status American Society of Anesthesiology Physical status 1,2

Exclusion Criteria:

* Ideal body weight >130% gastrointestinal disease prior administration of anti-emetics (24hr)

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-06; Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative nausea and vomiting | 24 hour postoperative

SECONDARY OUTCOMES:
incidence of postoperative nausea and vomiting | at immediate postoperative
incidence of postoperative nausea and vomiting | 6 hour postoperative
incidence of postoperative nausea and vomiting | 48 hour postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hee Kim, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou universiry hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No